CLINICAL TRIAL: NCT05405829
Title: Educational Intervention for Caregivers of the Elderly With Cognitive Impairment and Risk of Bronchial Aspiration, to Reduce Episodes of Pneumonia. A Randomized Clinical Trial.
Brief Title: Health Education to Caregivers to Reduce Aspiration Pneumonia
Acronym: HECGPN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Ana María Yuste Font, Principal Investigator, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INF-2018-08
Record Dates: First submitted 2022-05-18; First posted 2022-06-06 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Oropharyngeal Dysphagia; Pneumonia; Malnutrition
Keywords: Elderly, Swallowing Disorders, pneumonia, caregivers
MeSH Terms: conditions — Deglutition Disorders; Pneumonia; Malnutrition

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Conventional information received by caregivers. The speech therapist comes to the room to pass the Volume viscosity exploratory method test (V-VST) Test and after confirming dysphagia, informs the patient of the test result and delivers a booklet of recommendations.
  Interventions: Other: Health education
- Intervention group (Experimental): A 45-minute session, hygienic-dietary training, with visual support and work materials where three specific interventions are explained: textures for solids and liquids, safety postures to reduce the risk of bronchial aspiration, and oral hygiene. In addition, tools are offered to caregivers so that they can identify situations of anxiety and overload, as well as guidelines for social support.
  Interventions: Other: Health education

INTERVENTIONS:
Other: Health education — theoretical-practical hygienic-dietary training, with visual support and work materials where three specific interventions are explained: textures for solids and liquids, safety postures to reduce the risk of bronchial aspiration, and oral hygiene. In addition, tools are offered to caregivers so that they can identify situations of anxiety and overload, as well as guidelines for social support.

SUMMARY:
Randomized clinical study with a control group for assessing the decrease in the incidence of pneumonia, in a 12-month follow-up, in older people with cognitive impairment, risk of bronchial aspiration, risk of malnutrition and dependence to perform basic activities of daily living, through the design and implementation of an educational program. to the caregivers of these patients.

DETAILED DESCRIPTION:
Introduction: The number of people over 65 years of age is increasing, observing an older population worldwide. In the year 2050 there will be 2,000 million, this situation is due to medical and technological advances, in addition to the declining birth rate. People live longer, but there is also a higher incidence of chronic diseases, associated with age. Among them, neurodegenerative diseases stand out, due to the dependence they entail, as well as the risk of situations such as episodes of bronchial aspiration, which can cause pneumonia that will require hospital admissions, as well as the risk of malnutrition and dependence to carry out basic activities of daily life. .

Most of these patients are cared for at home by their caregivers, who, in addition to not knowing how to care for oropharyngeal dysphagia, the situation of prolonged fatigue can generate overload and anxiety for the caregiver.

Objective: To evaluate the decrease in the incidence of pneumonia, in a 12-month follow-up, in older adults with cognitive impairment, risk of bronchial aspiration, risk of malnutrition and dependence to carry out basic activities of daily living, through the design and implementation of a educational program. to the caregivers of these patients.

Methodology: A sequential exploratory mixed study will be carried out. For the design of the educational intervention, a descriptive qualitative study will be carried out with focus groups of caregivers and the recommendations of the Health Literacy model will be followed. To evaluate the efficacy of this intervention, a pre-post intervention randomized clinical trial with a control group will be carried out. The sample will be 178 couples made up of caregivers (formal or informal non-professional caregivers) and people over 65 who are in their care. The study will be carried out at the Parc Sanitari Per Virgili in Barcelona from May 2019 to March 2023. The main variables and study instruments are the incidence and admissions for pneumonia, as well as its delay in onset in older people, measured by Clinical history, cognitive impairment, measured with the Pfeiffer test, the risk of bronchial aspiration measured with the volumetric viscosity exploratory method test (V-VST), the risk of malnutrition measured with the Mini Nutritional Assessment short-form scale (MNA- SF). In addition to the anxiety and overload of their caregivers, measured with the Goldberg and Zarit scale.

ELIGIBILITY:
Patient inclusion criteria:

* People over 65 years of age, with cognitive impairment, evaluated with the Pfeiffer Test ≥ 3. With risk of bronchoaspiration, detected by the presence of oropharyngeal dysphagia and confirmed with the test (V-VST). Risk of malnutrition, evaluated with the MNA-SF test ≤ 11 and with dependency to perform the basic activities of daily living, with a Barthel index ≤ 61.
* Voluntary participation and signing the informed consent after being informed orally and in writing about the study, the patient or responsible relative.

Caregiver inclusion criteria:

* Voluntary participation and signing the informed consent after being informed orally and in writing about the study.

Patient exclusion criteria:

* Patients with a high degree of oropharyngeal dysphagia (that is, when they bronchoaspirate when administering 5 ml of pudding texture while performing the test (V-VST) to measure oropharyngeal dysphagia).
* Patients with delirium at the time of evaluation.
* Institutionalized patients, in residences or long stay.

Caregiver exclusion criteria:

* That the caregiver is not the usual one. This means that, at the time of the study, the patient is not cared for by the usual reference person. Therefore, the caregiver is present in a punctual and transitory situation.
* That patients or their caregivers do not understand the Catalan or Spanish language.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 178 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Variable: pneumonia. | At 12 months before entering the study; At 3 months before entering the study; At 3 months after entering the study; At 12 months after entering the study
  Qualitative variable, dichotomous (yes/no). Pneumonia is defined according to the International Classification of Diseases of the lungs (ICD 11), often caused by infection by bacteria, viruses, fungi or parasites, although not always. It is characterized by fever, chills, productive cough, chest pain, and dyspnea" (WHO 2022). Measured through self-prepared questionnaire and Clinical History.
Variable: time of onset of pneumonia. | At 3 months after entering the study; At 12 months after entering the study.
  Discrete quantitative variable. The elapsed time measured in months from the intervention to the appearance of the first pneumonia is considered.
Variable: Admission for pneumonia in the last year. | At 3 months after entering the study; At 12 months after entering the study.
  Qualitative, dichotomous variable (yes/no). Measured through own questionnaire.
Variable: Number of admissions for pneumonia in the last year. | At 12 months before entering the study; At 3 months before entering the study; At 3 months after entering the study; At 12 months after entering the study
  Discrete numerical quantitative variable. Measured through the Clinic History and own questionnaire.
Variable: Malnutrition risk. | At study entry; At 3 months after entering the study; At 12 months after entering the study
  Continuous quantitative variable. It is defined as "an unbalanced nutritional state resulting from insufficient nutrient intake to meet normal physiological requirements". Measured with Scale Mini Nutritional Assessment-Short Form (MNA-SF). Through the Clinic History and own questionnaire.
  Scale to assess malnutrition (maximum score of 14 points). 12-14 points: normal nutritional status; 8-11 points: risk of malnutrition; 0-7 points: malnutrition.
Variable: Cognitive impairment. | At study entry; At 3 months after entering the study; At 12 months after entering the study
  Discrete quantitative variable. Cognitive impairment is defined according to the Medical Subject Headings (MeSH) descriptor, as "the decrease or deterioration of mental and/or intellectual function". Measured with Pfeiffer test.
  Pfeiffer scale, It consists of 10 items. Between 0-2: it is considered normal; Between 3-4: mild cognitive impairment Between 5-7: moderate cognitive impairment; More than 8 errors: severe cognitive impairment.
Variable: Risk of Bronchoaspiration. | Before entering the study.
  Discrete quantitative variable. It is defined as "A type of pulmonary inflammation resulting from the aspiration of food, liquid, or gastric contents into the upper respiratory tract." Measured with the volume-viscosity swallow test (V-VST).
  Test performed to detect if there is aspiration due to dysphagia. The signs are: cough, decrease in basal oxygen saturation greater than 5%, change in tone of voice and/or alteration in efficacy such as insufficient lip seal, oral or pharyngeal residuals and fractional swallowing.
  The test consists of three textures (water, nectar and pudding) with three volumes (5 ml, 10 ml and 20 ml). It begins by administering (5ml of nectar texture), if any sign is found that compromises safety, it will not go to a higher volume or lower viscosity. It is concluded that there is no dysphagia when there are no signs of safety or altered efficacy at any time of the test.
Variable: Dependence to perform activities of daily living. | At study entry; At 3 months after entering the study; At 12 months after entering the study
  Ordinal quantitative variable. It is defined as the generic measure that assesses the patient's level of independence with respect to performing some basic activities of daily living. Measured by the Barthel Scale.
  It consists of 10 items, with different possible answers. Values from 0 points (total dependency) to 100 points (independent) < 20 total dependency; 20-35 severe dependency; 40-55 Moderate dependency; ≥ 60 mild dependency; 100 independent
Variable: Anxiety. | At study entry; At 3 months after entering the study; At 12 months after entering the study
  Qualitative variable. It is defined by the Medical Subject Headings (MeSH) "as feelings or emotions of fear, apprehension and impending disaster but not disabling as with anxiety disorders". It is measured by the Goldberg scale (Assessment of the Anxiety subscale) It consists of 10 items, its assessment ranges from 0 (no problem) to 10 points (severe anxiety) The cut-off points are 4 or more for the anxiety subscale
Variable: Burden. | At study entry; At 3 months after entering the study; At 12 months after entering the study
  Qualitative variable. It is defined as "as the caregiver's subjective experience of care demands, it is a multidimensional concept, with objective and subjective characteristics. The objective burden corresponds to the changes that the caregiver must make in various areas of life and the subjective burden refers to the emotional reactions to the demands of care". It is measured by the Zarit scale (Assessment of caregiver burden) It consists of 22 items, with five possible answers. Maximum score of 88 points. A score below 46 is usually considered indicative of "no overload", and a score above 56 of "severe overload".

SECONDARY OUTCOMES:
Variable: Level of Oropharyngeal Dysphagia. | At study entry; At 3 months after entering the study; At 12 months after entering the study
  Discrete quantitative variable. Coded as (level 1: severe dysphagia, novel 2: moderate-severe dysphagia, level 3: moderate dysphagia, level 4: mild-moderate dysphagia, novel 5: mild dysphagia, level 6: diet-modified functional swallowing, level 7, swallowing normal). It is defined as, "systematically rating the functional severity of dysphagia based on an objective assessment and making recommendations for the level of diet, level of independence, and type of nutrition" Measured with the Dysphagia Outcome and Severity Scale (DOSS).
Variable: Diet adherence | At 3 months after entering the study; At 12 months after entering the study
  Qualitative. Coded as (non-adherence, sequential, sporadic, partial or good). The WHO defines it as "the degree to which a patient's behavior, in relation to taking medication, following a diet or modifying lifestyle habits, corresponds to the recommendations agreed with the health professional" (World Health Organization). Health Organization 2003). Measured through the adherence questionnaire for dietary adaptations in dysphagia.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Gallart Fernández-Puebla, nursing, Study Director — Universitat Internacional de Catalunya; María Ángeles de Juan Pardo, nursing, Study Director — Universitat Internacional de Catalunya
Locations (1):
- Parc Sanitari Pere Virgili, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Boccardi V, Ruggiero C, Patriti A, Marano L. Diagnostic Assessment and Management of Dysphagia in Patients with Alzheimer's Disease. J Alzheimers Dis. 2016;50(4):947-55. doi: 10.3233/JAD-150931. PMID 26836016
- [Result] Nakamura K. [Aspiration pneumonia in elderly stroke patients in a convalescent rehabilitation ward: Risk factors and effects on recovery after stroke]. Nihon Ronen Igakkai Zasshi. 2020;57(1):45-52. doi: 10.3143/geriatrics.57.45. Japanese. PMID 32074560
- [Result] Hopwood J, Walker N, McDonagh L, Rait G, Walters K, Iliffe S, Ross J, Davies N. Internet-Based Interventions Aimed at Supporting Family Caregivers of People With Dementia: Systematic Review. J Med Internet Res. 2018 Jun 12;20(6):e216. doi: 10.2196/jmir.9548. PMID 29895512